CLINICAL TRIAL: NCT02835534
Title: The Efficacy and Safety of rhTNK-tPA in Comparison With Alteplase(Rt-PA) as Fibrinolytic Therapy of Acute ST Elevation Myocardial Infarction(STEMI): a Multi-center, Randomized, Open, Parallel, Non-inferiority, Active Controlled Trial
Brief Title: The Efficacy and Safety of rhTNK-tPA in Comparison With Alteplase(Rt-PA) as Fibrinolytic Therapy of Acute STEMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSPC Mingfule Pharmaceutical (Guangzhou) Co., Ltd. (Industry)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-2015-01
Record Dates: First submitted 2016-06-12; First posted 2016-07-18 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Acute ST Elevation Myocardial Infarction
Keywords: acute ST elevation myocardial infarction
MeSH Terms: interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhTNK-tPA (Experimental): rhTNK-tPA; Dose:16mg; Mode of admin: Single bolus Dose:50mg; Enoxaparin or unfractionated heparin for anticoagulant therapy, clopidogrel and aspirin for antiplatelet therapy before fibrinolytic therapy.
  Interventions: Drug: rhTNK-tPA
- rt-PA (Active Comparator): Drug:alteplase;Dose:50mg; Mode of admin: administered as an 8-mg initial IV bolus followed by an infusion of 42 mg over the next 90 minutes Enoxaparin or unfractionated heparin for anticoagulant therapy, clopidogrel and aspirin for antiplatelet therapy before fibrinolytic therapy.
  Interventions: Drug: alteplase

INTERVENTIONS:
Drug: rhTNK-tPA — Dose:16mg; Mode of admin: Single bolus Enoxaparin or unfractionated heparin for anticoagulant therapy, clopidogrel and aspirin for antiplatelet therapy before fibrinolytic therapy.
  Other Names: Recombinant Human TNK Tissue-type Plasminogen Activator
  Arms: rhTNK-tPA
Drug: alteplase — Dose:50mg; Mode of admin: administered as an 8-mg initial IV bolus followed by an infusion of 42 mg over the next 90 minutes Enoxaparin or unfractionated heparin for anticoagulant therapy, clopidogrel and aspirin for antiplatelet therapy before fibrinolytic therapy.
  Other Names: rt-PA
  Arms: rt-PA

SUMMARY:
This study is aiming to test the hypothesis that efficacy of rhTNK-tPA was not inferior to rt-PA with respect to the 30-day MACCE rates after fibrinolytic therapy for STEMI patients. It is a multicenter, randomized, open, parallel, active-controlled, non-inferiority trial.

DETAILED DESCRIPTION:
The study includes screening and baseline, randomization & intervention, in-hospital visit, at 30±3 days visit after fibrinolytic therapy.

Following an initial eligibility screening assessment, all eligible patients who have signed the informed consent will be randomly assigned by an interactive Web-based central system for fibrinolytic therapy with either rhTNK-tPA or rt-PA. The standard care should be given to all patients except for the study interventions.

Prior to fibrinolytic administration, enoxaparin (30-mg intravenous) or Un- Fractionated Heparin (maximum 4000U, intravenous) should be administered, combined with antiplatelet therapy consisted of both clopidogrel and aspirin in a 300-mg loading dose followed by routine dosage.

Successful reperfusion according to the clinical evidence (EKG) should be assessed after fibrinolytic therapy.TIMI flow should be assessed for those patients with 24 hours coronary angiography.

MACCE and bleeding events should be followed up and documented during the study until 30 days after fibrinolytic therap. An independent adjudication committee will judge the major endpoint events.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute STEMI（meet with both conditions）:

   * Ischemic chest pain ≥30mins in duration
   * ST elevation ≥0.1 mV in two or more limb ECG leads or ≥0.2 mV in two or more contiguous precordial leads
2. Onset of continuous ischemic symptoms of STEMI ≤6 hours prior to randomisation
3. Anticipated Delay to Performing Primary PCI >60mins，or time from hospital arrival to to balloon inflation >90mins
4. Signed Informed consent received prior to participation the study

Exclusion Criteria:

1. Non-ST-segment-elevation myocardial infarction or unstable angina
2. Reinfacrtion
3. Cardiacgenic shock
4. Suspected aortic dissection
5. New left bundle branch block in ECG
6. Absolute and relative contraindications for Fibrinolytic Therapy in STEMI(referred from 2015 China STEMI Management Guideline）：

   * Severe uncontrolled hypertension (unresponsive to emergency Therapy,BPs > 180 mmHg and/or BPd > 110 mmHg)
   * Any prior ICH,stroke with unknown cause, Ischemic stroke within 3 months
   * Known structural cerebral vascular lesion, malignant intracranial neoplasm
   * Active bleeding, or bleeding diathesis, active peptic ulcer
   * Significant closed-head or facial trauma within 3 months
   * Intracranial or intraspinal surgery within 2 months
   * Recent internal bleeding within 4 weeks
   * Major surgery within 3 weeks, or Traumatic
   * Prolonged cardiopulmonary resuscitation (>10 minutes)
   * Noncompressible vascular punctures within 2 weeks
   * Current use of anticoagulant therapy
7. Current or with a history of significant diseases：

   * Damage to the central nervous system
   * Severe renal or hepatic dysfunction, blood system diseases,
   * Present with cardiac rupture evidence
   * Acute pericarditis,Subacute bacterial endocarditis, Septic thrombophlebitis or occluded AV cannula at seriously infected site
   * Malignancy
   * High likelihood of left heart thrombus, e.g., mitral stenosis with atrial fibrillation
   * Diabetic hemorrhagic retinopathy or other hemorrhagic ophthalmic conditions
   * History of PCI or coronary artery bypass graft（CABG）within 1 month
8. Administration of fibrinlytic therapy prior to participation
9. Weight below 50 kg
10. Known current histroy of fall-down accident
11. Any other unfavourable conditions for participation：

    * Known participation in other clinical trials
    * Known to allergic to rhTNK-tPA or tPA or relevant vehicle
    * Pregnancy or lactation
    * Mental disorder
    * Present with any unsuitable conditions for participation or completion of the study at the discretion of their treating physician

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 818 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with TIMI grade 2 or 3 flow in the infarct-related artery after therapy (Limited to the subgroup for coronary angiography within 24 hours after therapy) | within 24 hours after therapy
  A patent IRA was defined as TIMI grade 2 or 3 flow on the angiogram

SECONDARY OUTCOMES:
The rate of MACCE (Major Adverse Cardiovascular and Cerebrovascular Events) | within 30 days after the start of fibrinolytic therapy
  MACCE composited of total death, non-fatal recurrent MI, non-fatal stroke (ischemic and Hemorrhage), PCI for failed reperfusion and PCI for reocclusion
The rate of successful reperfusion with clinical evidences | within 24 hours of fibrinolytic therapy
The in-hospital MACCE | during hospitalization (from the date of admission to the date of discharge, assessed up to 1 month)
The in-hospital and 30-day all-cause mortality | during hospitalization (from the date of admission to the date of discharge, assessed up to 1 month) and 30 days after the start of study interventions
The in-hospital and 30-day cardiac deaths | during hospitalization (from the date of admission to the date of discharge) and 30 days after the start of study interventions, assessed up to 1 month
The in-hospital recurrent MI | during hospitalization (from the date of admission to the date of discharge, assessed up to 1 month)
The 30-day revascularization | 30 days after the start of therapy
The in-hospital intracranial hemorrhage (ICH) | during hospitalization (from the date of admission to the date of discharge, assessed up to 1 month)
The in-hospital major GI bleeding events | during hospitalization (from the date of admission to the date of discharge, assessed up to 1 month)
The in-hospital total bleeding events | during hospitalization (from the date of admission to the date of discharge, assessed up to 1 month)

OTHER OUTCOMES:
The frequency and severity of AEs | during hospitalization (from the date of admission to the date of discharge, assessed up to 1 month)
Medical cost within the initial hospitalization | from the date of admission to the date of discharge, assessed up to 1 month
The frequency of re-hospitalizations and emergency room visits | at 30 days after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Shubin Qiaos, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital; Qin Yang, MD, Study Director — CSPC Mingfule Pharmaceutical (Guangzhou) Co., Ltd.
Locations (1):
- Guangzhou Recomgen Biotech Co., Ltd., Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao X, Zhu Y, Zhang Z, Tao G, Xu H, Cheng G, Gao W, Ma L, Qi L, Yan X, Wang H, Xia Q, Yang Y, Li W, Rong J, Wang L, Ding Y, Guo Q, Dang W, Yao C, Yang Q, Gao R, Wu Y, Qiao S. Tenecteplase versus alteplase in treatment of acute ST-segment elevation myocardial infarction: A randomized non-inferiority trial. Chin Med J (Engl). 2024 Feb 5;137(3):312-319. doi: 10.1097/CM9.0000000000002731. Epub 2023 Jun 2. PMID 37265385
- [Derived] Wang HB, Ji P, Zhao XS, Xu H, Yan XY, Yang Q, Yao C, Gao RL, Wu YF, Qiao SB. Recombinant human TNK tissue-type plasminogen activator (rhTNK-tPA) versus alteplase (rt-PA) as fibrinolytic therapy for acute ST-segment elevation myocardial infarction (China TNK STEMI): protocol for a randomised, controlled, non-inferiority trial. BMJ Open. 2017 Sep 18;7(9):e016838. doi: 10.1136/bmjopen-2017-016838. PMID 28928186